CLINICAL TRIAL: NCT03919136
Title: Accuracy of Non-Invasive Non-Oscillometric Blood Pressure Wrist Worn Measurement
Brief Title: Wrist Worn Blood Pressure Measurement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LiveMetric S.A. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB18-1281; NCT03911349 (obsolete NCT alias)
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Blood Pressure; Heart Failure; Advanced Heart Failure; Heart Failure，Congestive
Keywords: Heart Failure; Advanced Heart Failure; Blood Pressure; High Blood Pressure; Low Blood Pressure
MeSH Terms: conditions — Heart Failure; Hypertension; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Objective: Evaluation of the devices accuracy referenced to interventional (A-line) measurement.
  Interventions: Device: Wrist-worn measurement device (LiveMetric)

INTERVENTIONS:
Device: Wrist-worn measurement device (LiveMetric) — Evaluation of the wrist-worn measurement devices accuracy referenced to interventional (A-line) measurements.

SUMMARY:
In this study, the investigators are testing the accuracy of a wrist-worn measurement device by comparing its blood pressure measurement to arterial line (A-line) blood pressure monitors. The device is similar in style and fit to popular activity bands, but it is unique in that it measures blood pressure.

DETAILED DESCRIPTION:
LiveMetric has developed a wrist-worn measurement device intended for use as a standalone device, designed for measurement of intermittent blood pressure for individuals suffering from hypertension or other conditions where monitoring of blood pressure is of importance.

The wrist-worn measurement device is intended to be worn on the wrist for intermittent measurements of Blood pressure.

The use does not require any special action from the user apart from wearing the band on either their left or right wrist. The device applies no inflatable mechanics or moving parts. The wristband is watertight and can be worn as any type of bracelet all the time or most of the time.

The study will include subjects that are hospitalized in the ICU and/or any of the cardiology departments or affiliating units such as Cath lab, heart transplant unit, etc..) and are continually monitored by an intra-arterial blood pressure line (A-line). A medical professional will measure simultaneous non-invasive auscultatory readings to determine the lateral difference for later adjustment of calculation. A medical professional or a company representative accompanied by a medical professional will place the device on the opposite limb than the one having the A-line, providing the location of the placement has intact skin. During the measurement stage, BP values are simultaneously recorded from the reference invasive A-line and the wrist worn device.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a pre-existing intra-arterial blood pressure (A-Line) line for standard care
* Patients that are ≥18 years of age.

Exclusion Criteria:

* Body habitus that precludes patients from wearing a device on their wrist
* Subjects without normal palpable radial artery pulse, whether congenital, due to medical intervention, or otherwise
* Subjects with wrist circumference less than 155mm or greater than 210mm
* Subjects implanted with pacemaker, VAD's or other mechanical circulatory support device whether intracorporeal or extracorporeal
* Patients that do not have an intra-arterial blood pressure line.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an arterial line used for continuous blood pressure monitoring.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Non-Oscillometric Blood Pressure Wrist Worn Data Acquisition and Analysis | 2 years
  Measurements including systolic and diastolic pressures will be assessed and analyzed retrospectively according to the requirements of the standard (ISO 81060-2).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sayer, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - NYU School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sayer G, Piper G, Vorovich E, Raikhelkar J, Kim GH, Rodgers D, Shimbo D, Uriel N. Continuous Monitoring of Blood Pressure Using a Wrist-Worn Cuffless Device. Am J Hypertens. 2022 May 10;35(5):407-413. doi: 10.1093/ajh/hpac020. PMID 35171213